CLINICAL TRIAL: NCT01205126
Title: A Randomized, Double-Blind, Active Controlled, Multi-center Study to Investigate the Safety and Efficacy of OROS Hydromorphone HCl Once-daily Compared With Oxycodone HCL Controlled-release Twice Daily in Subjects With Cancer Pain
Brief Title: An Efficacy and Safety Study of Oral Osmotic Therapeutic System (OROS) Hydromorphone Hydrochloride (HCl) in Participants With Cancer Related Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR017437; 42801PAI3009
Record Dates: First submitted 2010-08-05; First posted 2010-09-20 (Estimated); Results first posted 2013-11-25 (Estimated); Last update posted 2014-02-03 (Estimated); Status verified 2013-12

CONDITIONS: Pain
Keywords: Pain; Hydromorphone hydrochloride; Oxycodone hydrochloride
MeSH Terms: conditions — Pain | interventions — Hydromorphone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- OROS Hydromorphone hydrochloride (HCl) (Experimental): OROS Hydromorphone HCl will be administered in dose of 8, 16, 24, and 32 milligram (mg), once daily for 2 to 8 days of titrationphase and 28 days of maintenance phase. Starting dose will be based on participant's previous daily opioid dose.
  Interventions: Drug: Hydromorphone HCl; Drug: Placebo
- Oxycodone HCl Controlled release (CR) (Active Comparator): Oxycodone HCl will be administered in dose of 10, 20, 30 and 40 mg, twice daily for 2 to 8 days of titrationphase and 28 days of maintenance phase. Starting dose will be based on participant's previous daily opioids dose.
  Interventions: Drug: Oxycodone HCl CR; Drug: Placebo

INTERVENTIONS:
Drug: Hydromorphone HCl — Hydromorphone HCl will be administered in dose of 8, 16, 24, and 32 milligram (mg), once daily for 2 to 8 days of Titration phase and 28 days of Maintenance phase. Starting dose will be based on participant's previous daily opioid dose.
  Arms: OROS Hydromorphone hydrochloride (HCl)
Drug: Oxycodone HCl CR — Oxycodone HCl will be administered in dose of 10, 20, 30 and 40 mg, twice daily for 2 to 8 days of titration phase and 28 days of maintenance phase. Starting dose will be based on participant's previous daily opioids dose.
  Arms: Oxycodone HCl Controlled release (CR)
Drug: Placebo — Placebo will be administered to the participants receiving hydromorphone HCl or oxycodone HCl CR along with the study treatment to maintain necessary blinding.

SUMMARY:
The purpose of this study is to compare the safety and efficacy of Oral Osmotic Therapeutic System (OROS) hydromorphone hydrochloride (HCl) with controlled-release oxycodone HCl in participants with cancer-related pain.

DETAILED DESCRIPTION:
This is a double-blind (a medical research study in which neither the researchers nor the participants know what treatment the participants is receiving), randomized (study drug is assigned by chance), multi-center (when more than one hospital or medical school team work on a medical research study), comparative, parallel-group (a clinical trial comparing the response in two or more groups of participants receiving different treatments) study of OROS hydromorphone HCl compared with oxycodone HCl controlled-release in participants with moderate to severe cancer (abnormal tissue that grows and spreads in the body until it kills) pain. The study will consist of 3 phases: a screening period (up to 14 days before randomization), a dose titration phase (up to 8 days), and a dose maintenance phase (28 days). The study visits will be scheduled at weekly intervals. Eligible participants will be randomly assigned to receive either hydromorphone HCl once daily or oxycodone HCl twice daily (placebo will be administered when necessary for blinding). During titration phase, dosage of hydromorphone HCl or oxycodone HCl will be adjusted upward or downward to achieve stable pain control. It can be from 2 days to 8 days. Participants who complete dose titration will enter into the dose maintenance phase and will receive study treatment for 28 consecutive days. Morphine hydrochloride will be given as rescue analgesic (drug used to control pain) medication for breakthrough pain during the study. Primarily efficacy will be evaluated by measuring change in the score of Brief Pain Inventory (BPI) questionnaire item 'worst pain' at end of maintenance period. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants receiving strong oral or transdermal (through the skin) opioid analgesics with inadequate control of moderate to severe (very serious, life threatening) cancer pain or who presented with cancer pain and will be eligible to move to Step 3 of the WHO analgesic ladder when receiving weak opioids
* Participants who require or are expected to require between 40 mg and 184 mg of oral morphine or morphine equivalents every 24 hours for the chronic management of cancer pain
* Participants who are reasonably expected to achieve a stable dose of opioid study medication during the study
* Participants who are not expected to start a course of chemotherapy, radiotherapy, targeted cancer therapy, hormone therapy or diphosphates therapy after enrolment into the study. If participants are receiving long-term treatment including hormone therapy, target cancer therapy and diphosphate, the treatment should be kept stable as much as possible from 2 weeks before randomization and up to the completion of the study, encompassing the titration and maintenance phases
* Female participants who are premenarchal, postmenopausal, or surgically sterile, abstinent or if sexually active, they must use a medically acceptable method of contraception and must be willing to continue to use the same method of contraception throughout the study

Exclusion Criteria:

* Participants with neuropathic pain or pain of unknown origin, or acute pain - Participants having pain only on movements
* Participants requiring other opioid analgesics (apart from morphine hydrochloride (HCl), in immediate release formulation, allowed as rescue medication for breakthrough pain)
* Participants with a recent history (within the previous 6 months) or current history of drug abuse or alcohol abuse
* Women of childbearing potential who were pregnant or lactating, seeking pregnancy or failing to use an adequate contraceptive method

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2009-12; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research and Development Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Locations (12):
- China (12):
  - Beijing
  - Chengdu
  - Fuzhou
  - Guangdong
  - Guangzhou
  - Hangzhou
  - Hefei
  - Nanchang
  - Nanning
  - Shanghai
  - Tianjin
  - Wuhan

RESULTS

PARTICIPANT FLOW:
Groups:
- Hydromorphone Hydrochloride (HCl): Osmotic Release Oral System (OROS) hydromorphone HCl was administered in dose of 8, 16, 24, and 32 milligram (mg), once daily for 2 to 8 days of titration phase and 28 days of maintenance phase. Starting dose was based on participant's previous daily opioid dose.
- Oxycodone HCl Controlled Release (CR): Oxycodone HCl was administered in dose of 10, 20, 30, and 40 mg, twice daily for 2 to 8 days of titration phase and 28 days of maintenance phase. Starting dose was based on participant's previous daily opioid dose.
Period: Titration Phase
Arm/Group | Hydromorphone Hydrochloride (HCl) | Oxycodone HCl Controlled Release (CR)
Started | 130 | 130
Completed | 107 | 111
Not Completed | 23 | 19
Not completed — Adverse Event | 5 | 3
Not completed — Withdrawal by Subject | 5 | 5
Not completed — Lost to Follow-up | 2 | 2
Not completed — No stable titration dose | 1 | 0
Not completed — More than maximum dosage required | 2 | 3
Not completed — Other | 8 | 6
Period: Between Titration & Maintenance Phase
Arm/Group | Hydromorphone Hydrochloride (HCl) | Oxycodone HCl Controlled Release (CR)
Started | 107 | 111
Completed | 107 | 107
Not Completed | 0 | 4
Not completed — Other | 0 | 4
Period: Maintenance Phase
Arm/Group | Hydromorphone Hydrochloride (HCl) | Oxycodone HCl Controlled Release (CR)
Started | 107 | 107
Completed | 70 | 67
Not Completed | 37 | 40
Not completed — Adverse Event | 3 | 7
Not completed — Death | 4 | 4
Not completed — More than the maximum dosage required | 5 | 5
Not completed — Prohibited drugs used | 1 | 0
Not completed — Other | 11 | 8
Not completed — Lost to Follow-up | 5 | 5
Not completed — Withdrawal by Subject | 8 | 11

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) population set included all the participants who were randomly assigned either of the 2 treatment groups and with at least 1 dose of medication administered during the titration phase and at least one assessment of efficacy.
Groups:
- Total: Total of all reporting groups
Arm/Group | Hydromorphone Hydrochloride (HCl) | Oxycodone HCl Controlled Release (CR) | Total
Number analyzed (Participants) | 125 | 123 | 248
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53.5 (10.86) | 52.7 (10.75) | 53.1 (10.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 43 | 86
  Male | 82 | 80 | 162

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Worst Pain in the Past 24 Hours Assessed by Brief Pain Inventory (BPI) Short Form Questionnaire Score at Day 29
Description: The BPI is questionnaire for evaluating the degree of pain severity and the impact of pain in performing daily routines. Change in worst pain in the past 24 hours in BPI score was reported. The total score ranges from 0 to 10, wherein 0 indicates no pain and 10 indicates pain as bad as participants could imagine.
Time Frame: Baseline and Day 29
Population: Per protocol set (PPS) included all randomly assigned participants who had completed all efficacy evaluations, and participants who prematurely discontinued the study due to lack of efficacy were also included. Redefined last observation carried forward (LOCF) was applied. Redefined LOCF is LOCF prior to over dose rescue medication.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Hydromorphone Hydrochloride (HCl) | Oxycodone HCl Controlled Release (CR)
Number analyzed (Participants) | 40 | 41
Units on a scale
  Baseline | 6.7 (1.80) | 6.9 (1.65)
  Change at Day 29 | -1.8 (2.79) | -1.8 (2.95)
Statistical Analysis 1: Comparison: Hydromorphone Hydrochloride (HCl) vs Oxycodone HCl Controlled Release (CR); Test type: Non-Inferiority or Equivalence — Non inferiority was demonstrated if upper bound of the 2-sided 95% CI was less than the non-inferiority margin of 1.5; p = 0.855, ANCOVA — P-value was calculated by ANCOVA model using Baseline as covariate for change at Day 29; Least square mean difference = -0.1, 95% CI 2-sided [-1.3 to 1.1], Standard Error of Mean 0.60

2. Secondary Outcome: Change From Baseline in Pain at Its Least, in the Past 24 Hours Assessed by BPI Short Form Questionnaire Score at Day 29
Description: The BPI is questionnaire for evaluating the degree of pain severity and the impact of pain in performing daily routines. Change in pain at its least, in the past 24 hours in BPI score was reported. The total score ranges from 0 to 10, wherein 0 indicates no pain and 10 indicates pain as bad as participants could imagine.
Time Frame: Baseline and Day 29
Population: The PPS included all randomly assigned participants who had completed all efficacy evaluations, have good compliance to the protocol without major protocol violations specified and who prematurely discontinued the study due to lack of efficacy were also included. Redefined LOCF was applied.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Hydromorphone Hydrochloride (HCl) | Oxycodone HCl Controlled Release (CR)
Number analyzed (Participants) | 40 | 41
Units on a scale
  Baseline | 2.4 (1.63) | 2.3 (1.37)
  Change at Day 29 | -0.8 (1.59) | -0.5 (2.20)
Statistical Analysis 1: Comparison: Hydromorphone Hydrochloride (HCl) vs Oxycodone HCl Controlled Release (CR); Test type: Non-Inferiority or Equivalence — Non inferiority was demonstrated if upper bound of the 2-sided 95% CI was less than the non-inferiority margin of 1.5; p = 0.615, ANCOVA; P-value was calculated by ANCOVA model using Baseline as covariate for change at Day 29; Least square mean difference = -0.2, 95% CI 2-sided [-1.0 to 0.6], Standard Error of Mean 0.39

3. Secondary Outcome: Change From Baseline in Average Pain, in the Past 24 Hours Assessed by BPI Short Form Questionnaire Score at Day 29
Description: The BPI is questionnaire for evaluating the degree of pain severity and the impact of pain in performing daily routines. Change in average pain in the past 24 hours, in BPI score was reported. The score ranges from 0 to 10 wherein, 0 indicates no pain and 10 indicates pain as bad as participants could imagine.
Time Frame: Baseline and Day 29
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Hydromorphone Hydrochloride (HCl) | Oxycodone HCl Controlled Release (CR)
Number analyzed (Participants) | 40 | 41
Units on a scale
  Baseline | 4.7 (1.35) | 4.7 (1.46)
  Change at Day 29 | -1.8 (1.98) | -1.4 (2.53)
Statistical Analysis 1: Comparison: Hydromorphone Hydrochloride (HCl) vs Oxycodone HCl Controlled Release (CR); Test type: Non-Inferiority or Equivalence — Non inferiority was demonstrated if upper bound of the 2-sided 95% CI was less than the non-inferiority margin of 1.5; p = 0.621, ANCOVA; P-value was calculated by ANCOVA model using Baseline as covariate for change at Day 29; Least square mean difference = -0.2, 95% CI 2-sided [-1.1 to 0.7], Standard Error of Mean 0.44

4. Secondary Outcome: Change From Baseline in Pain Right Now Assessed by BPI Short Form Questionnaire Score at Day 29
Description: The BPI is questionnaire for evaluating the degree of pain severity and the impact of pain in performing daily routines. Change in Pain Right now in BPI was reported. The score ranges from 0=no pain to 10=pain as bad as participants could imagine.
Time Frame: Baseline and Day 29
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Hydromorphone Hydrochloride (HCl) | Oxycodone HCl Controlled Release (CR)
Number analyzed (Participants) | 40 | 41
Units on a scale
  Baseline | 4.1 (2.09) | 4.1 (2.19)
  Change at Day 29 | -1.4 (2.60) | -1.4 (3.00)
Statistical Analysis 1: Comparison: Hydromorphone Hydrochloride (HCl) vs Oxycodone HCl Controlled Release (CR); Test type: Non-Inferiority or Equivalence — Non inferiority was demonstrated if upper bound of the 2-sided 95% CI was less than the non-inferiority margin of 1.5; p = 0.832, ANCOVA; P-value was calculated by ANCOVA model using Baseline as covariate for change at Day 29

5. Secondary Outcome: Change From Baseline in Pain Relief, in the Past 24 Hour Recorded Assessed by BPI Short Form Questionnaire at Day 29
Description: The BPI is questionnaire for evaluating the degree of pain severity and the impact of pain in performing daily routines. BPI comprises of total 9 items in total, and the 8th item consisting of 7 sub-items is a question asking the degree of disturbance due to pain. The score ranges from 0% to 100%, wherein 0% indicates no relief and 100% indicates complete relief.
Time Frame: Baseline and Day 29
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Hydromorphone Hydrochloride (HCl) | Oxycodone HCl Controlled Release (CR)
Number analyzed (Participants) | 40 | 41
Units on a scale
  Baseline | 48.8 (25.54) | 48.0 (23.05)
  Change at Day 29 | 15.8 (31.29) | 14.1 (32.01)
Statistical Analysis 1: Comparison: Hydromorphone Hydrochloride (HCl) vs Oxycodone HCl Controlled Release (CR); Test type: Non-Inferiority or Equivalence — Non inferiority was demonstrated if upper bound of the 2-sided 95% CI was less than the non-inferiority margin of 1.5; p = 0.304, ANCOVA; P-value was calculated by ANCOVA model using Baseline as covariate for change at Day 29

6. Secondary Outcome: Breakthrough Pain Medication (Rescue Medication) Doses Taken
Description: Any breakthrough pain medication taken during the overall study was reported. Morphine hydrochloride was used as a rescue medication in case of breakthrough pain.
Time Frame: Baseline up to Day 29
Population: The PPS included all randomly assigned participants who had completed all efficacy evaluations, have good compliance to the protocol without major protocol violations specified and who prematurely discontinued the study due to lack of efficacy. Redefined LOCF was applied. Here 'N' =number of participants who were evaluated for this outcome measure.
Measure: Mean (Standard Deviation); unit: Doses
Arm/Group | Hydromorphone Hydrochloride (HCl) | Oxycodone HCl Controlled Release (CR)
Number analyzed (Participants) | 36 | 40
Doses | 24.2 (24.41) | 29.3 (24.33)
Statistical Analysis 1: Comparison: Hydromorphone Hydrochloride (HCl) vs Oxycodone HCl Controlled Release (CR); Test type: Superiority or Other; p = 0.276, rank sum test, 2 sided

ADVERSE EVENTS:
Time Frame: Screening phase up to 30 days after last dose of study medication
Description: Safety set population included all the paricipants with at least 1 dose of study medication administered during the titration phase and at least one assessment of safety data.
Arm/Group | Hydromorphone Hydrochloride (HCl) | Oxycodone HCl Controlled Release (CR)
Serious Adverse Events (participants affected / at risk) | 11/128 | 18/126
Other Adverse Events (participants affected / at risk) | 102/128 | 107/126
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Hydromorphone Hydrochloride (HCl) (N=128) | Oxycodone HCl Controlled Release (CR) (N=126)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Bone marrow failure (Blood and lymphatic system disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 1 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Chest pain (General disorders) | 1 | 0
Death (General disorders) | 3 | 1
Disease progression (General disorders) | 0 | 1
Coma hepatic (Hepatobiliary disorders) | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 0 | 1
Jaundice (Hepatobiliary disorders) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Loss of consciousness (Nervous system disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 1 | 0
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Hydromorphone Hydrochloride (HCl) (N=128) | Oxycodone HCl Controlled Release (CR) (N=126)
Bone marrow failure (Blood and lymphatic system disorders) | 9 | 9
Anaemia (Blood and lymphatic system disorders) | 11 | 11
Abdominal discomfort (Gastrointestinal disorders) | 4 | 7
Abdominal distension (Gastrointestinal disorders) | 7 | 7
Constipation (Gastrointestinal disorders) | 43 | 45
Diarrhoea (Gastrointestinal disorders) | 12 | 9
Nausea (Gastrointestinal disorders) | 43 | 45
Vomiting (Gastrointestinal disorders) | 43 | 47
Asthenia (General disorders) | 11 | 9
Oedema peripheral (General disorders) | 11 | 6
Pyrexia (General disorders) | 24 | 27
Urinary tract infection (Infections and infestations) | 4 | 7
Neutrophil count decreased (Investigations) | 7 | 5
Platelet count decreased (Investigations) | 8 | 7
White blood cell count decreased (Investigations) | 13 | 17
Hypoproteinaemia (Metabolism and nutrition disorders) | 9 | 5
Decreased appetite (Metabolism and nutrition disorders) | 20 | 21
Dizziness (Nervous system disorders) | 21 | 22
Somnolence (Nervous system disorders) | 11 | 14
Chest discomfort (Respiratory, thoracic and mediastinal disorders) | 9 | 6
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3 | 8
Rash (Skin and subcutaneous tissue disorders) | 7 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less